CLINICAL TRIAL: NCT03890640
Title: Evaluation of the Accuracy of Real-time Ultrasound-assisted Thoracic Epidural Catheter Insertion: a Pilot Study
Brief Title: Ultrasound-assisted Thoracic Epidural Catheter Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jong Hyuk Lee, Clinical professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-0320
Record Dates: First submitted 2019-03-25; First posted 2019-03-26 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Abdominal Neoplasm; Thoracic Neoplasm
Keywords: Ultrasound; Thoracic epidural catheter insertion; Fluoroscopy
MeSH Terms: conditions — Abdominal Neoplasms; Thoracic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound-guided TECI (Experimental): After assessment of the epidural space using the loss of resistance technique with saline under ultrasound guidance, fluoroscopic views will be obtained to confirm which the catheter tip is located in the epidural space or not.
  Interventions: Procedure: Ultrasound-guided TECI

INTERVENTIONS:
Procedure: Ultrasound-guided TECI — When performing an ultrasound-guided thoracic epidural catheter insertion (TECI), an 18-gauge Tuohy needle will be used for interlaminar epidural access. All procedures will be performed with a paramedian approach under ultrasound-guidance and using the loss of resistance technique with saline. If the needle is deemed to be in the epidural space when the loss of resistance occurred, fluoroscopic views will be obtained to confirm which the catheter tip is located in the epidural space or not.

SUMMARY:
The aim of the present study is to access the success rate of ultrasound-guided thoracic epidural catheter insertion, using fluoroscopy.

DETAILED DESCRIPTION:
Thoracic epidural anesthesia has been associated with reduced acute postoperative pain for a wide variety of surgical procedures. It has also been associated with reductions in perioperative cardiac stress, chronic post-thoracotomy pain, and improvements in postoperative pulmonary function. Although a variety of methods can be used to confirm the position of the epidural needle in the epidural space, a blind technique and fluoroscopic guided approach are a widely used method. A thoracic epidural block is a relatively more difficult procedure than procedures used in other regions, because the spinous process of the thoracic vertebra is longer than that of the lumbar vertebra, and the area through which the needle can approach the epidural space is relatively smaller due to an acute angle and larger distance between the skin and the epidural space. Therefore, the success rate of thoracic epidural intervention is only about 68% under a blind technique due to inadequate position of the needle tip, misplacement, occlusion, and migration of the catheter.

Although fluoroscopic guided thoracic epidural intervention is the safest and most accurate method to identify the correct anatomical structures and confirm the epidural space with contrast medium, its use is limited because of the difficulty of using fluoroscope and the burden of radiation exposure. As the use of ultrasound has become popularized and universal, it has been widely used in regional anesthesia and analgesia, has continuously replaced the modality such as a blind technique and fluoroscopic guidance. Ultrasound-guided thoracic epidural catheter insertion was also recently investigated, and then it was conducted successfully in 15 cases of thoracic and upper abdominal surgery. Moreover, it showed several advantages including lowering the number of needle passes and increasing the success rate. However, it has not yet been studied how accurately the catheter is located in the thoracic epidural space during thoracic epidural catheter insertion using real-time ultrasound. Although it is possible to speculate the success of the thoracic epidural catheterization clinically, the identification of the location of the catheter is only possible under fluoroscopic guidance. Therefore, in the present study, we aimed to confirm the success rate of ultrasound-guided thoracic epidural catheter insertion, using fluoroscopy with contrast medium.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will undergo upper abdomen or thoracic surgery
* Scheduled for thoracic epidural catheter insertion
* 20 ≤ age <80
* When obtaining informed consent voluntarily

Exclusion Criteria:

* Allergy to local anesthetics and contrast dye, and steroid
* Use of anticoagulants or antiplatelet medication, coagulopathy
* Infection at the insertion site
* Neurological or psychiatric disorders
* Prior spine instrumentation
* Pregnancy

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-07-04 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Success rate of ultrasound-guided thoracic epidural catheter insertion | on the day of the procedure
  Confirmation success of ultrasound-guided thoracic epidural catheter insertion using fluoroscopic images; success means that the catheter tip is located in the epidural space.

SECONDARY OUTCOMES:
Number of skin punctures | on the day of the procedure
  complete needle withdrawal from the skin and reinsertion at a new location
Number of needle passes | on the day of the procedure
  First needle pass + additional needle passes (the needle returned to a plane perpendicular to the skin before reinsertion. Needle tip maneuvers toward the midline and cephalad were considered standard needle walking technique and were counted as a single pass)
First attempt success rate | on the day of the procedure
  only first needle pass and first skin puncture

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Hyuk Lee, MD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan medical center, Seoul, South Korea

REFERENCES:
- [Derived] Kim DH, Lee JH, Sim JH, Jeong W, Lee D, Kwon HM, Choi SS, Jeong SM. Real-time ultrasound-guided low thoracic epidural catheter placement: technical consideration and fluoroscopic evaluation. Reg Anesth Pain Med. 2021 Jun;46(6):512-517. doi: 10.1136/rapm-2021-102578. Epub 2021 Apr 23. PMID 33893174